CLINICAL TRIAL: NCT00006271
Title: Phase I/II Study of Neuroendocrine Dysfunction in Patients With Closed Head Injuries
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: National Center for Research Resources (NCRR) (NIH)
Collaborators: University of Texas (Other)
Other Study IDs: 199/15377; UTMB-96-422; UTMB-GCRC-453
Record Dates: First submitted 2000-09-11; First posted 2000-09-12 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 2003-12

CONDITIONS: Brain Injury
Keywords: brain injury; neurologic and psychiatric disorders; rare disease
MeSH Terms: conditions — Brain Injuries; Neurologic Manifestations; Mental Disorders; Rare Diseases

SUMMARY:
OBJECTIVES:

I. Determine the incidence of neuroendocrine dysfunction in patients with closed head injuries admitted to the Transitional Learning Community in Galveston, Texas, for rehabilitation.

DETAILED DESCRIPTION:
PROTOCOL OUTLINE: Phase I: Patients undergo fasting for urine and blood endocrine assessments. First morning urine is collected for measurement of 6-sulphatoxymelatonin (6-SMT). Following a medical history and a physical examination, patients undergo measurement of serum levels of free thyroxine, thyroid stimulating hormone (TSH), prolactin, insulin-like growth factor I (IGF-I), dehydroepiandrosterone-sulfate (DHEA-S), free and total testosterone (males only), and baseline growth hormone (GH). Female patients also provide a menstrual history and undergo screening for hypogonadism. Patients then undergo GH stimulation testing comprised of measurement of serum GH levels before and on 6 occasions during the 3 hours after receiving glucagon IV.

After eating, patients undergo adrenocorticotropic hormone stimulation testing comprised of measurement of serum cortisol levels before and at 45 minutes after receiving corticotropin IV.

Phase II: Beginning at noon on a different day, patients with any abnormal endocrine tests during phase I undergo 24 hour inpatient dynamic testing of the neuroendocrine system. Patients undergo GH stimulation testing comprised of measurement of serum GH levels before and on 4 occasions during the 2 hours after receiving levodopa. Patients also undergo concurrent thyrotropin releasing hormone (TRH) and gonadotropin releasing hormone (GnRH) stimulation testing comprised of measurement of serum TSH and luteinizing hormone (LH) levels before and at 15, 30, 60, and 90 minutes after receiving TRH and GnRH IV. Patients then undergo overnight metyrapone testing comprised of baseline measurement of serum 11-deoxycortisol and cortisol levels, followed by oral metyrapone with a snack, overnight fasting, and then remeasurement of serum 11-deoxycortisol and cortisol levels.

ELIGIBILITY:
PROTOCOL ENTRY CRITERIA:

--Disease Characteristics--

* Closed head injury that occurred at least 3 months ago
* Must be admitted to the Transitional Learning Community in Galveston, Texas, for rehabilitation

--Prior/Concurrent Therapy--

* No concurrent oral contraceptives or hormone replacement therapy

--Patient Characteristics--

* Mentally competent
* No legal guardian
* Not pregnant or nursing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100
Dates: Start 1997-01

CONTACTS AND LOCATIONS:
Overall Officials: Randall Urban, Study Chair — University of Texas
Locations (2):
- United States (2):
  - Transitional Learning Community, Galveston, Texas
  - University of Texas Medical Branch, Galveston, Texas